CLINICAL TRIAL: NCT01616654
Title: A Randomized, Multi-center, Investigator-blind, Vehicle- and Active-controlled, Phase 2 Study to Assess the Efficacy and Safety of Different Concentrations of CD5789 Cream Applied Once Daily in Subjects With Moderate to Severe Acne Vulgaris
Brief Title: Dose Range Study of CD5789 in Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18223
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene; tazarotene; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CD5789 25 mcg/g Cream (Experimental): Participants randomized in stratum 1, 2 and 3 were applied with 25 mcg/g CD5789 cream, once daily for 12 weeks.
  Interventions: Drug: CD5789 25 µg/g cream
- CD5789 50 mcg/g Cream (Experimental): Participants randomized in stratum 1, 2 and 3 were applied with 50 mcg/g CD5789 50 once daily for 12 weeks.
  Interventions: Drug: CD5789 50 µg/g cream
- CD5789 100 mcg/g Cream (Active Comparator): Participants randomized in stratum 1, 2 and 3 were applied with 100 mcg/g CD5789 cream, once daily for 12 weeks.
  Interventions: Drug: CD5789 100 µg/g cream
- Tazarotene 0.1% Gel (Placebo Comparator): Participants randomized in stratum 1 and 2 were applied with Tazarotene 0.1% Gel, once daily for 12 weeks.
  Interventions: Drug: Tazarotene 0.1% gel
- Vehicle Cream (Experimental): Participants randomized in stratum 1, 2 and 3 were applied with Vehicle Cream once daily for 12 weeks.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: CD5789 25 µg/g cream — CD5789 25 µg/g cream applied once daily
  Arms: CD5789 25 mcg/g Cream
Drug: CD5789 50 µg/g cream — CD5789 50 µg/g cream applied once daily
  Arms: CD5789 50 mcg/g Cream
Drug: CD5789 100 µg/g cream — CD5789 100 µg/g cream applied once daily
  Arms: CD5789 100 mcg/g Cream
Drug: Tazarotene 0.1% gel — Tazarotene 0.1% gel applied once daily
  Arms: Tazarotene 0.1% Gel
Drug: Vehicle cream — Vehicle cream applied once daily
  Arms: Vehicle Cream

SUMMARY:
To assess the efficacy and safety of different concentrations of CD5789 cream in participants with acne vulgaris for the purpose of dose identification.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant, 12 to 35 years old with the following characteristics:
* Facial acne severity grade of the following:

  * Stratum 1: IGA score of 3 or 4
  * Stratum 2: IGA score of 4
  * Stratum 3: IGA score of 3 or 4
* A minimum of 30 non-inflammatory lesions and fulfills the criteria of one of the following strata:

  * Stratum 1: A minimum of 20 but not more than 40 inflammatory lesions, and a maximum of one nodule on the face.
  * Stratum 2: More than 40 inflammatory lesions, and up to four nodules on the face.
  * Stratum 3: Participants of Japanese origin with at least 20 inflammatory lesions and up to four nodules on the face.

    * Note: Participants of Japanese origin will not be included in Stratum 1 or Stratum 2. Japanese origin is defined as all four grandparents were born in Japan.

Exclusion Criteria:

* The presence of severe forms of acne (acne conglobata, acne fulminans) or secondary acne form (chloracne, drug-induced acne, etc.)
* Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with the interpretation of the clinical trial results and/or put the participant at significant risk (according to the Investigator's judgment) if the participant participates in the clinical trial.
* Known or suspected allergies or sensitivities to any components of any of the study drugs.
* Current participation in any other clinical trial of a drug or device OR past participation within the 30 days prior to the Baseline visit.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 304 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2013-07-24 (Actual); Study Completion 2014-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, M.D., Study Director — Galderma R&D, Inc.
Locations (24):
- United States (24):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Parexel Early Phase, Glendale, California
  - Odyssey Medispa, Marina del Rey, California
  - Rady Children's Hospital, San Diego, California
  - FXM Research Corp Miami, Miami, Florida
  - FMX Research Miramar, Miramar, Florida
  - Meda Phase, Inc, Newnan, Georgia
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Dermatology Specialists PC, Louisville, Kentucky
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Skin Specialists, PC, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Zoe Drealos, MD, High Point, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Central Sooner Research, Norman, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Arlington Center for Dermatology, Arlington, Texas
  - Suzanne Bruce and Associates P.A. The Center for Skin Research, Houston, Texas
  - Stephen Miller MD, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in United States. A total of 422 participants were screened between 20 June 2012 to 01 May 2013. Of which, 118 were screen failures. Screen failures were mainly due to inclusion criteria not met. A total of 304 participants were randomized in the study.
Pre-assignment Details: Participants randomized were stratified according to ethnic origin, acne severity & number of lesions as: Stratum 1: Non-Japanese, Investigator's Global Assessment (IGA) of 3/4, >= 20 but <= 40 inflammatory and >=30 non-inflammatory lesions and <=1 nodule on face; Stratum 2: Non-Japanese, IGA of 4, >40 inflammatory & >= 30 non-inflammatory lesions and <=4 nodules on face; Stratum 3: Japanese origin, IGA of 3 or 4, >= 20 inflammatory & >= 30 non-inflammatory lesions & <= 4 nodules on face.
Groups:
- CD5789 25 mcg/g Cream: Participants randomized in stratum 1, 2 and 3 were applied with 25 microgram per gram (mcg/g) CD5789 cream, once daily for 12 weeks.
- CD5789 50 mcg/g Cream: Participants randomized in stratum 1, 2 and 3 were applied with 50 microgram per gram (mcg/g) CD5789 50 once daily for 12 weeks.
- CD5789 100 mcg/g Cream: Participants randomized in stratum 1, 2 and 3 were applied with 100 microgram per gram (mcg/g) CD5789 cream, once daily for 12 weeks.
Period: Overall Study
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | Vehicle Cream
Started | 61 | 61 | 60 | 61 | 61
Completed | 56 | 53 | 50 | 53 | 49
Not Completed | 5 | 8 | 10 | 8 | 12
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 3 | 1 | 5
Not completed — Protocol Violation | 0 | 5 | 2 | 4 | 4
Not completed — Lost to Follow-up | 1 | 0 | 3 | 2 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent to treat (ITT) population that included all participants who were randomized and to whom study drug was dispensed.
Groups:
- Total: Total of all reporting groups
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | Vehicle Cream | Total
Number analyzed (Participants) | 61 | 61 | 60 | 61 | 61 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.1 (5.26) | 18.2 (4.76) | 18.3 (5.59) | 18.3 (4.83) | 18.3 (4.84) | 18.2 (5.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 12 | 17 | 13 | 65
  Male | 46 | 53 | 48 | 44 | 48 | 239
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 0 | 2
  Asian | 0 | 2 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 8 | 12 | 13 | 49
  White | 52 | 51 | 52 | 47 | 47 | 249
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success Rate 1 (SR1)
Description: Success Rate 1 was defined as percentage of participants who achieved at least a two-point reduction in the Investigator Global Assessment (IGA) scale from baseline at week 12. Evaluation of acne was performed by the investigator based on the following 5 point scale: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, higher score indicated higher severity. All missing values were imputed by last observation carried forward (LOCF).
Time Frame: From Baseline at Week 12
Population: Analysis was performed on Intent to treat (ITT) population that included all subjects who were randomized and to whom study drug was dispensed.
Measure: Number; unit: percentage of participants
Groups:
- CD5789 Vehicle Cream: Participants randomized in stratum 1, 2 and 3 were applied with Vehicle Cream once daily for 12 weeks.
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | CD5789 Vehicle Cream
Number analyzed (Participants) | 61 | 61 | 60 | 61 | 61
percentage of participants | 29.51 | 32.79 | 26.67 | 32.79 | 16.39
Statistical Analysis 1: Comparison: CD5789 25 mcg/g Cream vs CD5789 Vehicle Cream; The 95% confidence interval on the difference between Vehicle and the specified treatment group success rates was based on normal approximation with continuity correction; Test type: Superiority; p = 0.096, Cochran-Mantel-Haenszel; Percentage difference = 13.115, 95% CI 2-sided [-3.266 to 29.495]
Statistical Analysis 2: Comparison: CD5789 50 mcg/g Cream vs CD5789 Vehicle Cream; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.040, Cochran-Mantel-Haenszel; Percentage difference = 16.393, 95% CI 2-sided [-0.249 to 33.036]
Statistical Analysis 3: Comparison: CD5789 100 mcg/g Cream vs CD5789 Vehicle Cream; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.184, Cochran-Mantel-Haenszel; Percentage difference = 10.273, 95% CI 2-sided [-5.923 to 26.470]
Statistical Analysis 4: Comparison: Tazarotene 0.1% Gel vs CD5789 Vehicle Cream; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.041, Cochran-Mantel-Haenszel; Percentage difference = 16.393, 95% CI 2-sided [-0.249 to 33.036]

2. Primary Outcome: Absolute Change From Baseline in Total Lesion Lesion Counts at Week 12 Using Last Observation Carried Forward (LOCF)
Description: The lesion counts were performed by the Investigator. Total lesion counts was the sum of inflammatory, non-inflammatory lesions and nodules. All missing values were imputed by LOCF.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | Vehicle Cream
Number analyzed (Participants) | 61 | 61 | 60 | 61 | 61
lesion count | -53.61 (8.314) | -54.75 (8.261) | -54.99 (8.296) | -59.84 (8.301) | -46.87 (7.934)
Statistical Analysis 1: Comparison: CD5789 25 mcg/g Cream vs Vehicle Cream; Analysis was performed using analysis of covariance (ANCOVA) with terms for treatment, stratum, and Baseline lesion count as covariate; Test type: Superiority; p = 0.108, ANCOVA; Percentage difference = -6.74, 95% CI 2-sided [-14.96 to 1.48]
Statistical Analysis 2: Comparison: CD5789 50 mcg/g Cream vs Vehicle Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.060, ANCOVA; Percentage difference = -7.88, 95% CI 2-sided [-16.11 to 0.34]
Statistical Analysis 3: Comparison: CD5789 100 mcg/g Cream vs Vehicle Cream; Analysis was performed using ANCOVA with terms for treatment, stratum, treatment stratum, and with Baseline lesion count as covariate; Test type: Superiority; p = 0.054, ANCOVA; Percentage difference = -8.11, 95% CI 2-sided [-16.35 to 0.13]
Statistical Analysis 4: Comparison: Tazarotene 0.1% Gel vs Vehicle Cream; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.002, ANCOVA; Percentage difference = -12.97, 95% CI 2-sided [-21.18 to -4.76]

3. Primary Outcome: Percentage Change From Baseline in Total Lesion Counts at Week 12 Using Last Observation Carried Forward (LOCF)
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | CD5789 Vehicle Cream
Number analyzed (Participants) | 61 | 61 | 60 | 61 | 61
percentage change | -47.59 (28.474) | -49.87 (24.731) | -50.72 (24.885) | -55.07 (26.295) | -40.48 (28.968)
Statistical Analysis 1: Comparison: CD5789 25 mcg/g Cream vs CD5789 Vehicle Cream; Test type: Superiority; p = 0.067, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: CD5789 50 mcg/g Cream vs CD5789 Vehicle Cream; Test type: Superiority; p = 0.054, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: CD5789 100 mcg/g Cream vs CD5789 Vehicle Cream; Test type: Superiority; p = 0.038, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Tazarotene 0.1% Gel vs CD5789 Vehicle Cream; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants With Success Rate 2 (SR2)
Description: Success Rate 2 (SR2) was defined as the percentage of participants rated "Clear" (Grade 0) or "Almost clear" (Grade 1) with at least a two-point reduction on the IGA scale from Baseline to Week 12. Evaluation of acne was performed by the investigator based on the following 5 point scale: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe, higher score indicated higher severity. All missing values were imputed by LOCF.
Time Frame: From Baseline to Week 12
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | Vehicle Cream
Number analyzed (Participants) | 61 | 61 | 60 | 61 | 61
percentage of participants | 13.11 | 14.75 | 16.67 | 21.31 | 8.20

5. Secondary Outcome: Absolute Change From Baseline in Inflammatory and Non-inflammatory Lesion Count up to Week 12 Using Last Observation Carried Forward (LOCF)
Description: The Inflammatory lesion count was the count of papules and pustules: papule was a small, solid elevation less than 1 cm in diameter, pustule was a small, circumscribed elevation of the skin that contains yellow-white exudate. The non-inflammatory lesion count was the count of open and closed comedones: Open comedone was a pigmented dilated pilosebaceous orifice (blackhead). Closed comedone was a tiny white papule (whitehead). All missing values were imputed by LOCF.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | CD5789 Vehicle Cream
Number analyzed (Participants) | 61 | 61 | 60 | 61 | 61
lesion count
  Inflammatory Lesions | -19.67 (14.874) | -21.11 (13.268) | -19.32 (11.566) | -21.03 (13.890) | -17.74 (15.073)
  Non-inflammatory Lesions | -24.30 (21.633) | -18.69 (12.895) | -23.70 (18.390) | -28.26 (26.346) | -17.70 (17.745)

6. Secondary Outcome: Percentage Change From Baseline in Inflammatory and Non-inflammatory Lesion Count up to Week 12 Using Last Observation Carried Forward (LOCF)
Description: The Inflammatory lesion count was the count of papules and pustules: papule was a small, solid elevation less than 1 cm in diameter, pustule was a small, circumscribed elevation of the skin that contains yellow-white exudate. The non-inflammatory lesion count was the count of open and closed comedones: Open comedone was a pigmented dilated pilosebaceous orifice (blackhead). Closed comedone was a tiny white papule (whitehead). All missing values were imputed by LOCF. Percent changes in lesion counts equals (Week 12 count minus Baseline count) divided by Baseline count multiplied by 100.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | CD5789 Vehicle Cream
Number analyzed (Participants) | 61 | 61 | 60 | 61 | 61
percentage change
  Inflammatory lesion count | -49.16 (35.711) | -53.14 (30.187) | -51.93 (27.255) | -53.09 (29.484) | -41.70 (35.898)
  Non-inflammatory lesion count | -46.34 (30.888) | -45.26 (29.331) | -49.57 (29.786) | -55.88 (28.913) | -38.20 (30.368)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) that occurred on or after the first dose of study medication through Week 14 Follow-up visit.
Description: The safety population was defined as the ITT population participants who applied/were administered the study drug(s) at least once.
Arm/Group | CD5789 25 mcg/g Cream | CD5789 50 mcg/g Cream | CD5789 100 mcg/g Cream | Tazarotene 0.1% Gel | CD5789 Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/60 | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 1/61 | 1/61 | 0/60 | 0/61 | 1/61
Other Adverse Events (participants affected / at risk) | 15/61 | 17/61 | 23/60 | 24/61 | 18/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD5789 25 mcg/g Cream (N=61) | CD5789 50 mcg/g Cream (N=61) | CD5789 100 mcg/g Cream (N=60) | Tazarotene 0.1% Gel (N=61) | CD5789 Vehicle Cream (N=61)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD5789 25 mcg/g Cream (N=61) | CD5789 50 mcg/g Cream (N=61) | CD5789 100 mcg/g Cream (N=60) | Tazarotene 0.1% Gel (N=61) | CD5789 Vehicle Cream (N=61)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1) | 5 (5) | 5 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 6 (6)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oppositional defiant disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide his draft of such publication to sponsor to review and approve at least 2 months prior to the date of intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.